CLINICAL TRIAL: NCT04391582
Title: Pediatric Burn Treatment Using Tilapia Skin as a Xenograft for Superficial-Partial Thickness Wounds: a Randomized Controlled Phase II Trial
Brief Title: Pediatric Burn Treatment Using Tilapia Skin as a Xenograft for Superficial-Partial Thickness Wounds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Responsible Party: Principal Investigator, Edmar Maciel Lima Júnior, Plastic Surgeon, Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pediatric Burn Tilapia Skin
Record Dates: First submitted 2020-04-30; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Burns
Keywords: Burns; Wounds and Injuries; Biocompatible Materials; Nile Tilapia; Oreochromis niloticus
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This was an open-label, monocentric, randomized phase II clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - Tilapia Skin (Experimental): After cleaning the lesion with tap water and 2% chlorhexidine gluconate, the tilapia skin was applied and covered with gauze and bandage.
  Interventions: Other: Tilapia skin
- Control - Silver sulfadiazine (Active Comparator): After cleaning the lesion with tap water and 2% chlorhexidine gluconate, a thin layer of silver sulfadiazine cream 1% was applied and covered with gauze and band
  Interventions: Drug: silver sulfadiazine cream 1%

INTERVENTIONS:
Other: Tilapia skin — After cleaning the lesion with tap water and 2% chlorhexidine gluconate, the tilapia skin was applied and covered with gauze and bandage. These dressings were changed only if the tilapia skin did not adhere properly to the wound bed
  Arms: Test - Tilapia Skin
Drug: silver sulfadiazine cream 1% — After cleaning the lesion with tap water and 2% chlorhexidine gluconate, a thin layer of silver sulfadiazine cream 1% was applied and covered with gauze and bandage. In these patients, the dressings were changed daily
  Arms: Control - Silver sulfadiazine

SUMMARY:
This study aims to evaluate the efficacy of Nile tilapia skin as a xenograft for the treatment of partial-thickness burn wounds in children.

DETAILED DESCRIPTION:
This is an open-label, monocentric, randomized phase II pilot study conducted in Fortaleza, Brazil. The study population consisted of 30 children between the ages of 2 and 12 years with superficial "partial-thickness" burns admitted less than 72 hours from the thermal injury. In the test group, the tilapia skin was applied. In the control group, a thin layer of silver sulfadiazine cream 1% was applied.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 2 and 12 years admitted to our institution with superficial partial thickness burns less than 72 hours from the thermal injury

Exclusion Criteria:

* Patients were excluded for a burn greater than 15% total body surface area (TBSA);
* Presence of a previous treatment for the current burn;
* Presence of a chemical or electrical burn;
* Presence of other significant diseases that could impact the volunteer's participation in the study;
* Presence of hypersensitivity to materials used in the study or to related compounds.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Complete burn wound healing | Day 11
  The number of days to complete burn wound healing (≥95% reepithelialization), calculated via clinical judgment from the consultant.
Assessment of pain via the Faces Pain Scale-Revised (FPS-R). | Day 11
  The pain evaluation via the FPS-R was performed by the patient himself or herself if aged 5 years or more, or by their caregiver in patients under 5 years of age. The scale consists of six faces, presented horizontally, that depict different degrees of pain, from "no pain" to "most pain possible". A numerical value from 0 to 10 is assigned to each face.
Assessment of pain via CONFORT-B scale. | Day 11
  The pain evaluation via CONFORT-B Scale was performed by the physician responsible and assessed the pain based in a behavioral that consisted in six factors: alertness, calmness/agitation, respiratory response (or crying), physical movement, muscle tone, and facial tension.Each factor was scored with values ranging between 1 and 5, generating scores between 6 and 30 points.
Assessment of pain via FLACCr scale. | Day 11
  The pain evaluation via FLACCr scale was performed by the physician responsible and answered five evaluation categories based on behavioral parameters with combined scores ranging from zero to ten (classified the scores as follows: zero to three (mild pain); four to six (moderate pain) and seven to ten (severe pain).

SECONDARY OUTCOMES:
Number of dressings performed. | Day 11
  In the test group, a dressing change was defined as the act of replacing the tilapia skin that did not adhere properly and/or replacing gauze and bandage that is full of exudate, after an evaluation of the dressing (performed every 48 hours). In the control group, a dressing change was defined as the daily act of cleaning the wound and reapplying the silver sulfadiazine cream 1%, which is then covered with new gauze and bandage.
Total amount of anesthetics and analgesics required throughout the treatment | Day 11
  To audit anesthetics and analgesics intake, nurses were trained to register on the patient's clinical record all analgesic and anesthetic medications used
Evaluation of burn improvement via the Clinical Global Impression Scale-Improvement (CGI-I). | Day 3, day 5, day 7, day 9 and day 11
  The CGI-I was evaluated by the physician responsible and answers the following question: "Compared to the patient's condition at admission to the project, this patient's condition is: 1 - very much improved since the initiation of treatment; 2 - much improved; 3 - minimally improved; 4 - no change from baseline; 5 - minimally worse; 6 - much worse; 7 - very much worse since the initiation of treatment"
Evaluation of burn severity via the Clinical Global Impression Scale- Severity (CGI-S). | Day 1, day 3, day 5, day 7, day 9 and day 11
  The CGI-I was evaluated by the physician responsible and answers the following question: "Compared to the patient's condition at admission to the project, this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."

CONTACTS AND LOCATIONS:
Locations (1):
- Burn Treatment Center, Dr. José Frota Institute, Fortaleza, Ceará, Brazil